CLINICAL TRIAL: NCT04133493
Title: A Multi-center, Randomized Controlled Clinical Trial Evaluating the Effect of Omega3 Wound Fish Skin Graft in the Treatment of Diabetic Foot Ulcers
Brief Title: Omega3 Wound Fish Skin Graft in the Treatment of DFUs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kerecis Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KS-0500
Record Dates: First submitted 2019-10-08; First posted 2019-10-21 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Diabetic Foot Ulcer
Keywords: fish skin graft; omega3 fatty acids
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled trial (RCT) with two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care Group (Placebo Comparator): Fibracol Dressing covered with gauze and wrapped with kerlix and wrap. Change 3Xper week
  Interventions: Device: Fibracol
- Intervention Group (Active Comparator): Kerecis affixed with steri-strips, cover with gauze and change one per week .
  Interventions: Device: Kerecis Omega3 Wound

INTERVENTIONS:
Device: Kerecis Omega3 Wound — The intervention group will receive, in addition, a fish skin graft (KerecisTM Omega3 Wound) secured with Steristrips, sutures or staples, covered with a nonadherent dressing (Adaptic, Systagenix, Yorkshire, UK or equivalent), the product bolstered down to the wound bed with a foam dressing (HydraFoam, DermaRite) and hydrogel as needed to retain adequate moisture balance and padded with stretch gauze and self adherent wrap as needed.
  The wound will be dressed by the site investigator 1 day a week.
  Arms: Intervention Group
Device: Fibracol — The Standard of Care Group will receive Fibracol covered with DSD. Change three times per week
  Arms: Standard of Care Group

SUMMARY:
The purpose of this clinical evaluation is to collect patient outcome data on a commercially available 510K FDA-approved product that is derived from minimal processing of Atlantic cod fish skin: KerecisTM Omega3 Wound.

In this trial, two groups of UT grade IA/1C diabetic foot ulcers (DFUs), full skin thickness or extending through the subcutaneous or fat layers but not into tendon, muscle, or bone will receive standard of care (SOC) treatment for their condition. Patients will be randomized to SOC treatment and a 510k FDA-approved collagen alginate dressing (Fibracol Plus) or SOC and KerecisTM Omega3 Wound. The primary endpoint is the percentage of index ulcers (the ulcers being treated in the study) healed at 12 weeks in which two groups that will be compared are SOC with Fibracol Plus or SOC with KerecisTM Omega3 Wound

DETAILED DESCRIPTION:
The study is a prospective, multi-center, parallel-group RCT designed to collect outcome data for the treatment of DFUs. The trial will be single blinded in regard to wound healing assessment (confirmation of wound healing will be overseen by an independent wound care adjudicator).

There are two arms in the study, both of which will receive standard of care (SOC): offloading of the DFU (CAM boots (Royce walker with diabetic inlay or equivalent) or total contact casting [TCC] if compliance issues or the subject's foot is too large for a CAM), appropriate sharp or surgical debridement. Patients cannot be on systemic antibiotics prior to randomization, infection management during treatment phase can include systemic antibiotics only in conjunction with debridement.

Arm 1 will receive, in addition, a fish skin graft (KerecisTM Omega3 Wound) secured with Steristrips, sutures or staples, covered with a nonadherent dressing (Adaptic, Systagenix, Yorkshire, UK or equivalent), the product bolstered down to the wound bed with a foam dressing (HydraFoam, DermaRite) and hydrogel as needed to retain adequate moisture balance and padded with stretch gauze and self adherent wrap as needed.

Arm 2 will receive a wound care covering comprising collagen alginate Fibracol plus dressing followed by a padded dressing comprised of 4x4 gauze pads, stretch gauze and self adherent wrap The wound will be dressed by patients or their caregivers at home 3 times a week and by the site investigator 1 day a week.

The study involves two phases: Screening and Treatment

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Presence of a DFU extending at least through the dermis but not into tendon, muscle, or bone, provided it is below the medial aspect of the malleolus (UT grade IA/IC; see Appendix A for definitions).
3. The index ulcer will be the largest ulcer if two or more eligible DFUs are present and will be the only one evaluated in the study. If other ulcerations are present on the same foot, they must be more than 2 cm distant from the index ulcer.
4. Index ulcer (i.e. current episode of ulceration) has been present for greater than 4 weeks prior to SV1 and less than 1 year, as of the date the subject consents for study.
5. Index ulcer is a minimum of 1.0 cm2 and a maximum of 25 cm2 at SV1 and TV1.
6. Adequate circulation to the affected foot as documented by a dorsal transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg, or an ankle brachial index (ABI) between 0.7 and 1.1 within 3 months of SV1, using the affected study extremity. As an alternative, arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle, or a toe brachial index (TBI) of > 0.6 is acceptable.
7. The target ulcer has been offloaded for at least 14 days prior to randomization.
8. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers or abstinence) during the course of the study and undergo pregnancy tests.
9. Subject understands and is willing to participate in the clinical study and can comply with weekly visits

Exclusion Criteria:

1. Index ulcer(s) deemed by the investigator to be caused by a medical condition other than diabetes.
2. Index ulcer, in the opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a carcinoma of the ulcer.
3. Index ulcer on the heel
4. Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within 1-month prior to first SV1, or who receive such medications during the screening period or who are anticipated to require such medications during the course of the study.
5. Subjects on any investigational drug(s) or therapeutic device(s) within 30 days preceding SV1.
6. Subjects who have received a biomedical or topical growth factor for their wound within the previous 30 days.
7. History of radiation at the ulcer site (regardless of time since last radiation treatment).
8. Index ulcer has been previously treated or will need to be treated with any prohibited therapies. (See Section 7.3 of this protocol for a list of prohibited medications and therapies).
9. Subject has a known history of poor adherence with medical treatment.
10. Osteomyelitis or bone infection of the affected foot as verified by x-ray within 30 days prior to randomization. (In the event of an ambiguous diagnosis, the Principal Investigator will make the final decision).
11. Subject is pregnant or breast-feeding.
12. Presence of diabetes with poor metabolic control as documented with an HbA1c >12.0 within 90 days of randomization.
13. Subjects with end stage renal disease as evidenced by a serum creatinine ≥ 3.0 mg/dL within 6 months of randomization.
14. Index ulcer has reduced in area by 20% or more after 14 days of SOC from SV1 to the TV1/randomization visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Wound Healing | 12 weeks
  A comparison of the proportion of index ulcers healed at 12 weeks. This is a "Yes/No" assessment The wounds can either be "healed" or "not healed".

SECONDARY OUTCOMES:
Time to Heal | 12 weeks
  Measurement of total time to healing
PAR | 12 weeks
  Percent Area Reducation at 12 weeks
Pain reduction: visual analogue scale (VAS) | 12 weeks
  measured by visual analogue scale (VAS). The subject will be asked to indicate a numerical value that best represents the pain intensity at the index ulcer site on a scale of 0 (minimum value) to 10 (maximum value). The number 0 represents "no pain" the number 5 represents "moderate pain" and the number 10 represents "worst possible pain"

OTHER OUTCOMES:
Histology assessment from biopsies | 12weeks
  Changes in histology features

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Lullove, DPM, Principal Investigator — Eric J. Lullove DPM, PA; Gunnar Johannsson, PhD, Study Director — Kerecis Ltd.; John Lantis, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (5):
- United States (5):
  - Eric J. Lullove DPM, PA, Coconut Creek, Florida
  - Village Podiatry Centers - Smyrna (Allen Raphael, DPM), Smyrna, Georgia
  - Christopher Winters, DPM, Carmel, Indiana
  - Brock Liden, DPM, Circleville, Ohio
  - Bert J. Altmanshofer, DPM, Duncansville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: An Economic Evaluation of the Impact, Cost, and Medicare Policy Implications of Chronic Nonhealing Wounds. — https://www.ncbi.nlm.nih.gov/pubmed/29304937
- See also: Cost-of-illness studies in chronic ulcers: a systematic review. — https://www.ncbi.nlm.nih.gov/pubmed/28379102
- See also: Healing of diabetic neuropathic foot ulcers receiving standard treatment. A meta-analysis. — https://www.ncbi.nlm.nih.gov/pubmed/10332667
- See also: Predictors of lower-extremity amputation in patients with an infected diabetic foot ulcer. — https://www.ncbi.nlm.nih.gov/pubmed/25665817
- See also: A Prospective, Postmarket, Compassionate Clinical Evaluation of a Novel Acellular Fish-skin Graft Which Contains Omega-3 Fatty Acids for the Closure of Hard-to-heal Lower Extremity Chronic Ulcers. — https://www.ncbi.nlm.nih.gov/pubmed/27071138
- See also: Regenerative and Antibacterial Properties of Acellular Fish Skin Grafts and Human Amnion/Chorion Membrane: Implications for Tissue Preservation in Combat Casualty Care. — https://www.ncbi.nlm.nih.gov/pubmed/28291503
- See also: A novel bioactivity of omega-3 polyunsaturated fatty acids and their ester derivatives. — https://www.ncbi.nlm.nih.gov/pubmed/20331795
- See also: The antibacterial properties of docosahexaenoic omega-3 fatty acid against the cystic fibrosis multiresistant pathogen Burkholderia cenocepacia. — https://www.ncbi.nlm.nih.gov/pubmed/22150831
- See also: The marine Omega3 wound matrix for treatment of complicated wounds A multicenter experience report — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6096721/
- See also: Treatment of diabetic foot wounds with acellular fish skin graft rich in omega-3: a prospective evaluation. — https://www.ncbi.nlm.nih.gov/pubmed/30767649
- See also: Healing rate and autoimmune safety of full-thickness wounds treated with fish skin acellular dermal matrix versus porcine small-intestine submucosa: a noninferiority study. — https://www.ncbi.nlm.nih.gov/pubmed/25759413
- See also: Fish-Skin Grafts Compared to Human Amnion/Chorion Membrane Allografts: A Double-Blind, Prospective, Randomized, Clinical Trial of Acute Wound Healing. — https://www.ncbi.nlm.nih.gov/pubmed/31509319
- See also: A cross-sectional validation study of using NERDS and STONEES to assess bacterial burden. — https://www.ncbi.nlm.nih.gov/pubmed/19717855
- See also: Determination of ideal PtcO2 measurement time in evaluation of hypoxic wound patients. — https://www.ncbi.nlm.nih.gov/pubmed/18351126